CLINICAL TRIAL: NCT03057171
Title: A Study on the Gastrointestinal Disease and Helicobacter Pylori Controlled Long Non-coding RNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0146
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Helicobacter Pylori Infection; Gastric Ulcer; Duodenal Ulcer; Stomach Cancer
Keywords: Helicobacter pylori; long non-coding RNA; THRIL; PACER; cagA
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EGD, forcep biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Gastric ulcer: patients who will undergo EGD for gastric ulcer
- Duodenal ulcer: patients who will undergo EGD for duodenal ulcer
- Stomach cancer: patients who will undergo EGD for stomach cance
- health individuals: patients who will undergo screening EGD

SUMMARY:
Helicobacter pylori (H.pylori) is a major human pathogenic bacterium in gastric mucosa which is linked to the development of gastritis, peptic ulcer disease, mucosa-associated lymphoid tissue lymphoma and gastric cancer. However the regulatory mechanism of H.pylori-induced immune response is not clear. Long non-coding RNA (lncRNA) has recently emerged as key post-transcriptional regulators of gene expression, differentiation. The investigators had a preliminary results which THRIL (TNFα and hnRNPL related immunoregulatory lincRNA) and PACER(p50-associated COX-2 extragenic RNA) played a potential role in H.pylori induced inflammatory cascade. However, there wasn't a previous study about expression of THRIL, PACER in a human tissue. Therefore, the investigators aimed to evaluate the expression of THRIL, PACER in patients with gastrointestinal disease according to H.pylori infection.

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old
2. Patients with gastric ulcer
3. Patients with duodenal ulcer
4. Patients with stomach cancer
5. Patients with gastrointestinal discomfort symptoms

Exclusion Criteria:

1. Patients who has done helicobacter pylori eradication
2. Patients who has undergone gastrectomy
3. Patients who has undergone endoscopic submucosal dissection
4. Patients with active upper gastrointestinal bleeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal disease associated with H.pylori infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Expression of THRIL, PACER | Within 2 weeks after EGD
  Expression of THRIL, PACER according to Helicobacter pylori infection by Real-time aRT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No